CLINICAL TRIAL: NCT04150978
Title: Effectiveness of Early Enteral Feeding With High Protein Formulas Versus Oligomeric Formula Versus 5% Dextrose Solution in Clinical Improvement and Malnutrition Prevention of Intensive Care Unit Patients. A Quasi-Experimental Design
Brief Title: High Protein Formula on Enteral Feeding in Clinical Improvement and Malnutrition at Intensive Care Unit Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3110191419
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Critically Ill; Intensive Care Unit
Keywords: High Protein Polymeric Feeding; APACHE II Score; SOFA Score; NUTRIC Score; Critical Illness; Intensive Care Unit; Oligomeric Protein Feeding
MeSH Terms: conditions — Critical Illness | interventions — Peptamen; Glucose

STUDY DESIGN:
Intervention Model Description: Within 24-48 hours, Intensive care patients are allocated into three treatment, Enteral High-Protein Formulas, Oligomeric Formula, and 5% Dextrose Solution as control
Who Masked: Investigator
Masking Description: The investigator is blinded from any information regarding the treatment allocation of participants during the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 5% Dextrose (Active Comparator): the parenteral formulation as prescribed by the intensive care specialist
  Interventions: Drug: 5% Dextrose
- High Protein Polymeric Formula (Experimental): Procedure :
  1. The daily calorie and protein prescriptions were calculated from standard recommendations (calories 25-30 kcal/kg/d, proteins 1.2-2 g/kg/d)
  2. Administered as boluses via a nasogastric tube. A total of 5 aliquots were administered at 4-hourly intervals in a daily feeding period of 24 hours, with the participant positioned 30° head-up.
  Interventions: Other: High Protein Polymeric Formula
- Oligomeric Formula (Experimental): Similar to the High Protein Polymeric Formula Procedure
  Interventions: Other: Oligomeric Formula

INTERVENTIONS:
Other: High Protein Polymeric Formula — Component: 22.4% protein from total calorie Preparation of Peptisol: 5 spoons of Peptisol powder diluted in 200 ml warm water to have 250 ml Peptisol (equal to 250 kcal). Given as written in the group descriptions
  Other Names: Peptisol
  Arms: High Protein Polymeric Formula
Other: Oligomeric Formula — Component: Component: 22.4% protein from total calorie Preparation: 5 spoons of Peptamen powder diluted in 165 ml warm water to have 200 ml Peptamen (equal to 200 kcal). Given as written in the group descriptions
  Other Names: Peptamen
  Arms: Oligomeric Formula
Drug: 5% Dextrose — 500 ml of 5% Dextrose administered to a peripheral vein.
  Other Names: D5
  Arms: 5% Dextrose

SUMMARY:
Effectiveness of Early Enteral Feeding With High Protein Polymeric Formula Versus Oligomeric Formula Versus 5% Dextrose Solution in Clinical Improvement and Malnutrition on Intensive Care Unit Patients

Background :

Critically ill patients are physiologically unstable, often have complex hypermetabolic responses to trauma. These patients are facing a high risk of death, multi-organ failure, and prolonged ventilator use. Nutrition is one of therapy for critical illness, however, patients often experience malnutrition caused by disease severity, delays in feeding, and miscalculation of calorie needs, therefore, appropriate management of enteral feeding formula should be done in preventing malnutrition and improve clinical outcome during intensive treatment.

Objective:

This study aims to evaluate clinical improvement and malnutrition in critically ill participants under two different early enteral feeding formulas versus parenteral feeding

Methodology :

A three-arm randomized trial is performed (parenteral (5% Dextrose), and enteral high-protein polymeric formula, and oligomeric formula.) at the Intensive Care Unit in Wahidin Sudirohusodo Hospital, Makassar, Indonesia. The enteral feedings are given through a nasogastric tube within 24-48 hours after intensive care unit (ICU) admission as well as the parenteral group. A meticulous record of the calories and protein of intake is maintained for 3 days follow up including clinical parameters. The changes between pre and post-intervention of clinical parameters and nutrition scoring are assessed as the outcome of the intervention

Hypothesis :

Enteral feeding with High Protein Formula provides a better clinical outcome and less malnutrition event in comparison to 5% Dextrose and Oligomeric Formula

DETAILED DESCRIPTION:
Procedure :

1. All patients admitted to the Intensive care unit will undergo eligibility screening
2. Baseline assessments will be performed to eligible participants upon the first 24 hours including :

   1. anthropometric data (age, gender, height (participant in the supine position), ideal body weight (IBW), Mid-Upper-Arm Circumference (MUAC), and primary admission diagnosis (Traumatic Brain Injury/TBI or non-TBI).
   2. Laboratory assessment including platelets, white blood cells, lymphocytes, serum creatinine levels, blood urea nitrogen (BUN) levels, albumin, serum potassium levels, serum sodium levels, serum pH, the partial pressure of carbon dioxide, and partial pressure of oxygen (PO2)
   3. Scoring of Severity-of-illness using the laboratory parameters and clinical parameters under SOFA, APACHE II Score and NUTRIC score elements
3. The allocation of the participants is performed through simple randomization with the masking of the investigator.
4. the intervention will be done according to the protocol of each arm.
5. Measurement of outcomes according to the time frame by the intensive care and nutritionist team.
6. Data analysis including descriptive statistics and outcome analysis using paired t-test or Wilcoxon signed-rank test. Differences in mean values between the 3 groups are compared using the ANOVA or Kruskal-Wallis test. A p-value <0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

- stable hemodynamic values

Exclusion Criteria:

* gastrointestinal resection
* contraindications for enteral feeding
* history of diabetes or chronic kidney disease
* given parenteral nutrition
* had severe intolerance for enteral nutrition or formula
* gastric residual volume > 250 ml/4 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-07-07 (Actual)

PRIMARY OUTCOMES:
Nutrition Risk in the Critically Ill (NUTRIC) Score | 3 days after intervention initiated
  The Nutrition Risk in the Critically Ill (NUTRIC) Score is designed to quantify the risk of critically ill patients developing adverse events that may be modified by aggressive nutrition therapy ranging from 1-10. A score between 0-5 indicates a low malnutrition risk and 6 above means the patient is associated with worse clinical outcomes (mortality, ventilation) and the most likely to benefit from aggressive nutrition therapy.

OTHER OUTCOMES:
Sequential Organ Failure Assessment Score (SOFA) Score | Upon admission to Intensive Care Unit and 3 days after intervention
  The sequential organ failure assessment score (SOFA score) is a clinical scoring to determine the extent of a person's organ function or rate of failure during a stay in an intensive care unit (ICU) including the assessment of respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. The elements including PaO2/FiO2 (mmHg), Glasgow Coma Scale, Mean arterial pressure OR administration of vasopressors required, Bilirubin Level, Platelets, and Creatinine (mg/dl) [μmol/L] (or urine output). Each domain has scale from 0-4, with a total score for all domains is 24. Higher number indicates severe organ failure.
Acute Physiology, Age, Chronic Health Evaluation (APACHE) Score II | Upon admission to Intensive Care Unit and 3 days after intervention
  Acute Physiology, Age, Chronic Health Evaluation (APACHE) Score II is an ICU-scoring system to measure the risk and severity of the disease, including :
  AaDO2 or PaO2 (depending on FiO2) Temperature (rectal) Mean arterial pressure pH arterial Heart rate Respiratory rate Sodium (serum) Potassium (serum) Creatinine Hematocrit White blood cell count Glasgow Coma Scale. An integer score from 0 to 71 is computed based on measurements above; higher scores correspond to more severe disease and a higher risk of death

CONTACTS AND LOCATIONS:
Overall Officials: Agussalim Bukhari, MD, Ph.D, Principal Investigator — Hasanuddin University
Locations (1):
- Wahidin Sudirohusodo General Hospital, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berg A, Rooyackers O, Bellander BM, Wernerman J. Whole body protein kinetics during hypocaloric and normocaloric feeding in critically ill patients. Crit Care. 2013 Jul 24;17(4):R158. doi: 10.1186/cc12837. PMID 23883571
- [Background] Biolo G, Tipton KD, Klein S, Wolfe RR. An abundant supply of amino acids enhances the metabolic effect of exercise on muscle protein. Am J Physiol. 1997 Jul;273(1 Pt 1):E122-9. doi: 10.1152/ajpendo.1997.273.1.E122. PMID 9252488
- [Background] Biolo G, Grimble G, Preiser JC, Leverve X, Jolliet P, Planas M, Roth E, Wernerman J, Pichard C; European Society of Intensive Care Medicine Working Group on Nutrition and Metabolism. Position paper of the ESICM Working Group on Nutrition and Metabolism. Metabolic basis of nutrition in intensive care unit patients: ten critical questions. Intensive Care Med. 2002 Nov;28(11):1512-20. doi: 10.1007/s00134-002-1512-2. Epub 2002 Oct 1. PMID 12415440
- [Background] Dungan KM, Braithwaite SS, Preiser JC. Stress hyperglycaemia. Lancet. 2009 May 23;373(9677):1798-807. doi: 10.1016/S0140-6736(09)60553-5. PMID 19465235
- [Background] Higgins PA, Daly BJ, Lipson AR, Guo SE. Assessing nutritional status in chronically critically ill adult patients. Am J Crit Care. 2006 Mar;15(2):166-76; quiz 177. PMID 16501136
- [Background] Kim H, Stotts NA, Froelicher ES, Engler MM, Porter C. Enteral nutritional intake in adult korean intensive care patients. Am J Crit Care. 2013 Mar;22(2):126-35. doi: 10.4037/ajcc2013629. PMID 23455862
- [Background] Lena D, Kalfon P, Preiser JC, Ichai C. Glycemic control in the intensive care unit and during the postoperative period. Anesthesiology. 2011 Feb;114(2):438-44. doi: 10.1097/ALN.0b013e3182078843. No abstract available. PMID 21245729
- [Background] Löfgren E, Md. 2015. Early enteral nutrition compared to outcome in critically ill trauma patients at a level one trauma centre. S Afr J Clin Nutr;28(2):70-76
- [Background] Marik PE, Bellomo R. Stress hyperglycemia: an essential survival response! Crit Care. 2013 Mar 6;17(2):305. doi: 10.1186/cc12514. PMID 23470218
- [Background] de Souza Menezes F, Leite HP, Koch Nogueira PC. Malnutrition as an independent predictor of clinical outcome in critically ill children. Nutrition. 2012 Mar;28(3):267-70. doi: 10.1016/j.nut.2011.05.015. Epub 2011 Aug 27. PMID 21872433
- [Background] Mowery NT, Dortch MJ, Dossett LA, Norris PR, Diaz JJ Jr, Morris JA Jr, May AK. Insulin resistance despite tight glucose control is associated with mortality in critically ill surgical patients. J Intensive Care Med. 2009 Jul-Aug;24(4):242-51. doi: 10.1177/0885066609335663. Epub 2009 Jul 17. PMID 19617231
- [Background] Soeters MR, Soeters PB. The evolutionary benefit of insulin resistance. Clin Nutr. 2012 Dec;31(6):1002-7. doi: 10.1016/j.clnu.2012.05.011. Epub 2012 Jun 7. PMID 22682085